CLINICAL TRIAL: NCT06402110
Title: Femoral Triangle Block Versus Adductor Canal Block for Analgesia After Arthroscopic Anterior Cruciate Ligament Reconstruction: A Randomized Trial
Brief Title: Femoral Triangle Block Versus Adductor Canal Block in Arthroscopic Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MS559/4/24
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Femoral Triangle Block; Adductor Canal Block; Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral Triangle Block (FTB) Group (Experimental): Patients will receive femoral triangle block (FTB) at the end of surgery.
  Interventions: Other: Femoral Triangle Block
- Adductor Canal Block (ACB) Group (Experimental): Patients will receive adductor canal block (ACB) at the end of surgery.
  Interventions: Other: Adductor Canal Block

INTERVENTIONS:
Other: Femoral Triangle Block — Patients will receive femoral triangle block (FTB) at the end of surgery. The probe will be positioned at the level where the medial border of the sartorius muscle intersects the medial border of the adductor longus muscle, a block needle advanced in an in-plane technique into femoral triangle. After negative aspiration, 2ml of saline will be injected to confirm the needle tip position close to the femoral artery then injection of 15ml of bupivacaine 0.25% will be performed.
  Arms: Femoral Triangle Block (FTB) Group
Other: Adductor Canal Block — Patients will receive adductor canal block (ACB) at the end of surgery. The probe will be positioned at the point midway between the anterior superior iliac spine and the upper pole of the patella. The adductor canal will be located as a hyperechoic structure beneath the Sartorius muscle and a block needle advanced in an in-plane technique toward the target nerve after negative aspiration, 2ml of saline will be injected into adductor canal to confirm the block needle tip within it, the block needle will be advanced with the guidance of ultrasound in an in-plane technique and 15ml bupivacaine 0.25% will be injected.
  Arms: Adductor Canal Block (ACB) Group

SUMMARY:
The aim of this study is to compare the postoperative analgesic effect of femoral triangle block (FTB) and adductor canal block (ACB)after arthroscopic anterior cruciate ligament (ACL) reconstruction.

DETAILED DESCRIPTION:
The number of patients undergoing arthroscopic anterior cruciate ligament (ACL) reconstruction has risen over the past decade. ACL reconstruction is associated with moderate to severe postoperative pain leading to hypertension, tachycardia, increased O2 demand, and myocardial stress.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I and II.
* Undergoing elective arthroscopic Anterior Cruciate Ligament (ACL) reconstruction.

Exclusion Criteria:

* Revisional surgery.
* Body mass index (BMI) >35kg/m2.
* Coagulopathy.
* Infection at site of intervention.
* Hypersensitive to the study drugs.
* Chronic analgesic use.
* Neuromuscular disease.
* Drug abuse.
* Cognitive impairment.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-04-27 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of 3 mg morphine IV will be given if the Numeric Rating Scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4. NRS will be assessed at 2, 4, 6, 12, and 24h postoperatively

SECONDARY OUTCOMES:
Time of 1st rescue analgesia | 24 hours postoperatively
  Postoperatively, all patients will receive paracetamol 1gm/6h and diclofenac sodium 75mg I.M/12h as regular analgesia. Rescue analgesia of 3 mg morphine IV will be given if the Numeric Rating Scale (NRS) > 3 to be repeated after 30 min if pain persists until the NRS < 4. NRS will be assessed at 2, 4, 6, 12, and 24h postoperatively.
Pain score using Numeric Rating Scale (NRS) | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) (0 represents "no pain" while 10 represents "the worst pain imaginable"). It will be assessed at 2, 4, 6, 12, and 24h postoperatively.
Quadriceps strength | 24 hours postoperatively
  Quadriceps strength will be assessed at 2, 4, 6, 12, and 24h postoperatively. The criteria for evaluation of quadriceps strength are as follow: I (no contraction), II (have contraction, but cannot move joint), III (can move joint, but cannot resist gravity), IV (can resist gravity, but cannot bear substantial resistance), V (can bear a certain intensity of resistance), and VI (can bear full resistance).
Patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.